



### **Study Protocol Template (non CTIMP Interventional)**

Study Title: Emergency Cerclage in Twin Pregnancies at Imminent Risk of Preterm Birth: an Open-Label Randomised Controlled Trial

ENCIRCLE Trial (Emergency Cerclage in Twin Pregnancies at Imminent Risk of Preterm Birth: an Open-Label Randomised Controlled Trial)

**Sponsor's Project Number:** 17.004 **REC Reference Number:** 17/EE/0040

**IRAS ID: 222216** 

Version 1.7 15th May 2018

### **CHIEF INVESTIGATOR (CI):**

#### Dr Asma Khalil

Consultant in Obstetrics and Fetal Medicine
Fetal Medicine Unit
4th Floor Lanesborough Wing
St George's University Hospitals NHS Foundation Trust
Tooting
London
SW17 0QT

Phone: 0208 725 0071/07917400164

**Email:** akhalil@sgul.ac.uk **Fax:** +44 20 8725 0079

SPONSOR: St George's University Hospitals NHS Foundation Trust





#### **SPONSOR REPRESENTATIVE:**

Name Nadia Azzouzi

Address: St George's Joint Research Enterprise Office

Hunter Wing, Ground Floor,

Cranmer Terrace, London SW17 ORE

**Phone:** 02082666488

Email: <u>nazzouzi@squl.ac.uk</u>

**Fax:** 020 8725 0794

**Funding Source**: The trial is partially funded by the Twins And Mutiple Births Association (TAMBA).

Information in this protocol is confidential and should not be disclosed, other than to those directly involved in the execution or the ethical review of the study, without written authorisation from St George's Joint Research & Enterprise Office (JREO) or its affiliates.





#### **UK Collaborators:**

# Public and Patient Involvement Representative Mr Keith Reed

Chief Executive
Twins and Multiple Birth Association (TAMBA)
Manor House
Manor Park
Church Hill
Aldershot

### Prof. Baskaran Thilaganathan

Fetal Medicine Unit St George's NHS Foundation Trust Blackshaw Road Tooting LONDON SW17 0RE

Email: <a href="mailto:basky@pobox.com">basky@pobox.com</a>

### **Miss Rosemary Townsend**

Fetal Medicine Unit St George's NHS Foundation Trust Blackshaw Road Tooting LONDON SW17 0RE

Email: rosemary.townsend1@nhs.net

#### Mr Amar Bhide

Fetal Medicine Unit St George's NHS Foundation Trust Blackshaw Road Tooting LONDON SW17 0RE abhide@squl.ac.uk

### Mr Austin Ugwumadu

Fetal Medicine Unit St George's NHS Foundation Trust Blackshaw Road Tooting





LONDON SW17 0RE Austin.Ugwumadu@stgeorges.nhs.uk

### Mr George Attilakos

Fetal Medicine Unit University College Hospital 235 Euston Road Bloomsbury LONDON NW1 2BU

Email: George.Attilakos@uclh.nhs.uk

#### Miss Melanie Griffin

Senior Clinical fellow and Clinical Lecturer in Obstetrics and Gynaecology St Michael's Hospital Southwell Street Bristol BS2 8EG

Email: Melanie.Griffin@UHBristol.nhs.uk

### **Prof. Alan Cameron**

Queen Elizabeth University Hospital 1345 Govan Road Glasgow G51 4TF

Email: Alan.cameron@clinmed.gla.ac.uk

### Ms Christina Yu

Queen Charlotte's Hospital Du Cane Road Shepherd's Bush LONDON W12 0HS

Email: Christina.Yu@imperial.nhs.uk

### **Prof. Christoph Lees**

Queen Charlotte's Hospital Du Cane Road Shepherd's Bush LONDON W12 0HS

Email: <a href="mailto:christoph.Lees@imperial.nhs.uk">christoph.Lees@imperial.nhs.uk</a>





#### Mr Andrew Breeze

Leeds Teaching Hospitals NHS Trust Great George Street Leeds LS1 3EX

Email: andrewbreeze@nhs.net

### **Ms Catriona Monaghan**

Regional Fetal Medicine Unit Royal Jubilee Maternity Hospital 274 Grosvenor Road Belfast BT12 6BA

Email: <a href="mailto:camonaghan@doctors.org.uk">camonaghan@doctors.org.uk</a>

#### Ms Ferha Saeed

Newham University Hospital Glen Road Plaistow LONDON E13 8SL

Email: Ferha.Saeed@bartshealth.nhs.uk

### Ms Luxmi Velauthar

Newham University Hospital Glen Road Plaistow LONDON E13 8SL

Email: Luxmimalar.Velauthar@bartshealth.nhs.uk

### **Professor Shakila Thangaratinam**

Women's Health Research Unit
Barts and the London School of Medicine and Dentistry
Yvonne Carter Building
58 Turner Street
Whitechapel
LONDON
D1 2AB

Email: s.thangaratinam@qmul.ac.uk

### **Dr Andrew Sharp**

Liverpool Womens Hospital

Crown Street





Liverpool L8 7SS

Email: a.sharp@liverpool.ac.uk

### **Professor Zarko Alfirevic**

Liverpool Womens Hospital Crown Street Liverpool L8 7SS

Email: zarko@liv.ac.uk

#### **Dr Simon Grant**

North Bristol NHS Trust Southmead Hospital Southmead Road Westbury-on-Trym Bristol BS10 5NB

Email: <a href="mailto:simon.grant@nbt.nhs.uk">simon.grant@nbt.nhs.uk</a>

### **Dr Amanda Bellis**

Royal Preston Hospital Sharoe Green Lane North Fulwood Preston PR2 9HT

Email: Amanda.Bellis@lthtr.nhs.uk

### **Dr Penelope McParland**

Leicester Royal Infirmary Infirmary Square Leicester LE1 5WW

Email: Penelope.mcparland@uhl-tr.nhs.uk

### **Dr Tommy Mousa**

Leicester Royal Infirmary Infirmary Square Leicester LE1 5WW

Email: tommy.mousa@uhl-tr.nhs.uk

### Dr Latha Vinyakarao

Poole Hospital NHS Trust Longfleet Road Poole BH15 2JB





Email: <u>Latha.Vinayakarao@poole.nhs.uk</u>

### Dr Sharmila Sivarajan

Surrey and Sussex NHS Trust East Surrey Hospital Canada Avenue Redhill RH1 5RH

Email: <a href="mailto:sharmila.sivarajan@sash.nhs.uk">sharmila.sivarajan@sash.nhs.uk</a>

#### **Miss Renata Hutt**

Royal Surrey County Hospital Egerton Road Guildford GU2 7XX

Email: renata.hutt@gmail.com

### Miss Kasia Gajewska-Knapik

Cambridge University Hospitals The Rosie Hospital Robinson Way Cambridge CB2 0SW

Email: kgajewska@doctors.org.uk

### Mr Hiran Samarage

Northwick Park Watford Road Harrow Middlesex HA1 3UJ

Email: hiran.samarage@nhs.net

Miss Surabhi Nanda St Thomases Hospital Westminster Bridge Road Lambeth LONDON SE1 7EH

TBC Lewisham Hospital Lewisham High Street





### LONDON SE13 6LH

### Non-UK Collaborators:

### Prof. Dr. Liesbeth Lewi

University Hospitals Leuven Fetal Medicine Unit Herestraat 49 3000 Leuven, Belgium

Tel: +32 16 34 28 62

Email: <u>liesbeth.lewi@uzleuven.be</u>

#### Prof. Dr. Yves Ville

University Clinic Necker-Enfants Malades Department of Gynaecology and Obstetric 149 Rue de Sevres, 75015 Paris, France

E-mail: <a href="mailto:ville.yves@gmail.com">ville.yves@gmail.com</a>
Phone: +33 144381710

### Prof. Dr. Eduardo Gratacos

Hospital Clínic Sede Maternitat Fetal Medicine Center C/ Sabino de Arana, 1, 08028

Barcelona, Spain

E-mail: <u>Gratacos@clinic.ub.es</u> Phone: +34 932279931

### Dr. Greg Ryan

Mount Sinai Hospital Joseph and Wolf Lebovic Health Complex 1001-522 University Avenue Toronto, Ontario, Canada

E-mail: <a href="mailto:gryan@mtsinai.on.ca">gryan@mtsinai.on.ca</a>
Phone: +1 4165868403

### Prof. Dr. Jon Hyett

RPA Women and Babies, Royal Prince Alfred Hospital Missenden Road Camperdown NSW 2050, Australia

E-mail: jon.hyett@sswahs.nsw.gov.au

Phone: +61 295158887

### Prof. Dr. Christoph Berg





Universitätsklinikum Bonn Sigmund-Freud Strasse 25 53105 Bonn, Germany

E-mail: <a href="mailto:christoph.berg@ukb.uni-bonn.de">christoph.berg@ukb.uni-bonn.de</a>

Phone: +49 228-28714728

#### Dr. Romain Favre

**CMCO-SIHCUS** 

Schiltigheim/Strasbourg, France E-mail: <a href="mailto:romain.favre3@orange.fr">romain.favre3@orange.fr</a>

Phone: +33 388628329 - 0621720553

### Dr. Peter Lindgren

Karolinska University Hospital S 141 86 Stockholm, Sweden

E-mail: <a href="mailto:peter.lindgren@karolinska.se">peter.lindgren@karolinska.se</a>

Phone: +46 706092923

#### Dr. Francisca Molina

San Cecilio University Hospital

C/ Dr Oloriz, 16.18012 Granada, Spain

E-mail: fsoniamolina@gmail.com

### Dr. Roland Zimmerman

University Hospital Zurich

Frauenklinikstrasse 10, Zürich, Switzerland

E-mail: roland.zimmermann@usz.ch

Phone: +41 442555101

### Dr. Nicola Persico

Ospedale Maggiore Policlinico Via della Commenda 12 20122 Milan, Italy

E-mail: Nicola.persico@gmail.com

### Prof. Dr. Dick Oepkes

Leiden University Medical Center Department of Obstetrics, K-06-35 P.O. Box 9600, 2300RC Leiden, The Netherlands

Tel: +31 715 26 28 96 Email: <u>d.oepkes@lumc.at</u>

### **Dr. Enrico Lopiore**





Leiden University Medical Center Department of Pediatrics, Division of Neonatology P.O Box 9600, 2300 RC Leiden The Netherlands

Email: e.lopriore@lumc.nl

#### **Prof. Tiran Dias**

Faculty of Medicine University of Kelaniya Colombo North Teaching Hospital Ragama, Colombo

Email: thiran dias@yahoo.com

### **Prof. Rogelio Cruz Martinez**

Unit for Investigation of Fetal Medicine and Surgery Hospital de Especialidades del Nino y la Mujer de Queretaro Universidad Nacional Autónoma de México (UNAM) Querétaro. México

Email: rcruz@medicinafetalmexico.com

E-mail: mn193@leicester.ac.uk

### **Dr Minu Nath**

Senior Biomedical Statistician

Department of Cardiovascular Sciences

University of Leicester

British Heart Foundation Cardiovascular Research Centre

Glenfield General Hospital, Groby Road,

Leicester, LE3 9QP, UK

### **Statement**

The Chief Investigator (CI) and the Sponsor representative have discussed this protocol version. The investigators agree to perform the investigations and to abide by this protocol except where departures from it are mutually agreed in writing.

The Investigator agrees to conduct the trial in compliance with the protocol, GCP, the Data Protection Act (1998), the Trust Information Governance Policy (or other local equivalent), the Research Governance Framework (2005 2<sup>nd</sup> Edition), the Sponsor's SOPs, and other regulatory requirements as appropriate.

This protocol has been written in accordance to the Sponsor's procedure identified as: JREOSOP0039 "Protocol Design" and is intended for use at UK sites only

| Chief Investigator | Signature | Date |
|---|---|---|
| Asma Khalil | | |
| Consultant in Obstetrics and Fetal Medicine | MM | 20.11.2016 |
| St George's University Hospitals NHS Foundation Trust | | |

**Acknowledgements and Protocol contributories** 

### **Contents**

| 1 | List | of abbreviations | 14 |
|---|---|---|---|
| 2 | Rol | es and Responsibilities | 15 |
| 3 | Stu | dy synopsis | 16 |
| 4 | Bac | ckground | 11 |
| 5 | Stu | dy objectives | 13 |
| | 5.1 | Primary objective | 13 |
| | 5.2 | Secondary objectives | 13 |
| 6 | Tria | al design | 13 |
| 7 | Par | ticipation selection criteria | 13 |
| | 7.1 | Inclusion criteria | 22 |
| | 7.2 | Exclusion criteria | 22 |
| 8 | Par | ticipant Recruitment process | 22 |
| 9 | Stu | dy procedures | 23 |
| | 9.1 | Informed consent | 23 |
| | 9.2 | Randomisation procedure | 24 |
| | 9.3 | Discontinuation/withdrawal of participants and stopping rules | 24 |
| | 9.5 | Participant transfers | 25 |
| | 9.4 | Lost to Follow up | 25 |
| | 9.5 | Definition of the End of Trial | 25 |
| 1( | ) Stu | dy Procedures | 25 |
| | 10.1 | Measurement of cervical length | 23 |
| | 10.2 | Screening for infections | 25 |
| | 10.3 | Baseline assessment | 26 |
| | 10.4 | Intervention | 24 |
| | 10.5 | Follow-up visits | 26 |
| | 10.6 | Data collection | 26 |
| | 10.7 | Summary flow chart of study assessments | 26 |
| 1 | 1 Stu | dy Timeline | 27 |
| 12 | | ety Events | 27 |
| | 12.1 | Definitions | 27 |
| | 12.2 | Recording Adverse Events (AEs) | |
| | 12.3 | Investigator Responsibilities relating to Safety Reporting | 20 |
| | 12.4 | Notification of deaths | 20 |
| 1 | 3 Dat | a management and quality assurance | 20 |
| | 13.1 | Confidentiality | |
| | 13.2 | Data collection tool | 20 |
| | 13.3 | Incidental Findings | 21 |
| | 13.4 | Data handling and analysis | |
| | | hiving arrangements | |
| 1 | 5 Sta | tistical design | |
| | 15.1 | Endpoints | |
| | 15. | | 21 |
| | 15. | 1.2 Secondary endpoints | 21 |

| 15.2 | Sample size calculation | 22 |
|--------|------------------------------------------------------------|----|
| 15.3 | · | |
| 16 Et | hics and Research Governance requirements | |
| 16.1 | Annual Progress Reports (APRs) | |
| 16.2 | | |
| 16.3 | Direct access to source data | 32 |
| 17 Fii | nance | 32 |
| 18 Ins | surance and indemnity | 33 |
| 19 IP | and development policy | 33 |
| 22 Pu | ıblication policy | 33 |
| 20.1 | Before the official completion of the Trial | 33 |
| 20.2 | Up to 180 days after the official completion of the Trial | 34 |
| 20.3 | Beyond 180 days after the official completion of the Trial | 34 |
| 21 St | atement of Compliance | 34 |
| 22 Li | st of Protocol appendices | 35 |
| 23 R | eferences | 35 |

### 1 List of abbreviations

CI Chief Investigator
CRF Case Report Form
GCP Good Clinical Practice
ICF Informed Consent Form
ISF Investigator Site File

NHS R&D National Health Service Research & Development

PI Principal Investigator

PIS Participant Information Sheet **RCT** Randomised Controlled Trial Research Ethics Committee **REC** SDV Source Document Verification SOP Standard Operating Procedure SSA Site Specific Assessment **Trial Management Group TMG TSC Trial Steering Committee** 

### 2 Roles and Responsibilities

### **CHIEF INVESTIGATOR (CI):**

### Dr Asma Khalil

Consultant in Obstetrics and Fetal Medicine
Fetal Medicine Unit
4th Floor Lanesborough Wing
St George's University Hospitals NHS Foundation Trust
Tooting
London
SW17 0QT

Phone: 07917400164/0208 725 0071

**Email:** akhalil@sgul.ac.uk **Fax:** +44 20 8725 0079

SPONSOR: St George's University Hospitals NHS Foundation Trust

### **SPONSOR REPRESENTATIVE:**

Name Nadia Azzouzi

Address: St George's Joint Research Enterprise Office

Hunter Wing, Ground Floor,

Cranmer Terrace, London SW17 ORE

**Phone:** 02082666488

Email: nazzouzi@squl.ac.uk

**Fax:** 020 8725 0794

# 3 Study synopsis

| Brief title: | ENCIRCLE trial |
|---|---|
| Official title: | Emergency Cerclage in Twin Pregnancies at Imminent Risk of Preterm Birth: an Open-Label Randomised Controlled Trial |
| Sponsor reference number: | 17.0004 |
| Public database identifier | TBC |
| Study design | Pilot randomised controlled trial |
| Study<br>Population/disease<br>condition | <ul> <li>2 groups</li> <li>Twin pregnancies between 14 – 26 weeks' gestation presenting with an open cervix</li> <li>Monochorionic twin pregnancies complicated by twin-to-twin transfusion syndrome (TTTS) treated by Laser surgery between 16+0 and 26+0 weeks' gestation in whom a short cervix (&lt;15mm) is identified</li> </ul> |
| Eligibility criteria: | <ul> <li>Inclusion criteria:</li> <li>Twin pregnancies presenting with an open cervix between 14 and 26 weeks of gestation, OR</li> <li>Twin pregnancies complicated by TTTS treated by Laser surgery between 16+0 and 26+0 weeks' gestation in whom a short cervix (&lt;15mm) is identified.</li> <li>Age &gt;18 years</li> <li>Informed consent</li> <li>Exclusion criteria: <ul> <li>Cervical dilatation ≥5cm</li> <li>Amniotic membranes prolapsed beyond external os into the vagina, unable to visualise cervical tissue</li> <li>Preterm premature rupture of the membranes (PPROM) at the time of diagnosis of dilated cervix</li> <li>Major fetal malformations unrelated to TTTS</li> <li>Intrauterine death of one or both fetuses</li> <li>Symptoms or signs of threatened imminent delivery, e.g. painful regular uterine contractions, active vaginal bleeding, history of ruptured membranes</li> </ul> </li> <li>Suspected chorioamnionitis [based on maternal uterine tenderness, a temperature of 38°C or greater, significant leucocytosis (&gt;15,000 x 10<sup>6</sup>/L) or elevated C-reactive protein (&gt;15 mg/L), or maternal tachycardia].</li> </ul> |

| | Placenta praevia |
|---|---|
| | Monochorionic monoamniotic twin pregnancies |
| | Prophylactic cervical cerclage |
| | Women who are not able to give valid consent, e.g. unconscious or severely ill |
| | <ul> <li>Mental health disorder which impairs the ability to give<br/>fully informed consent</li> </ul> |
| | Women under the age of 18 years |
| | Higher order multiple pregnancies |
| Target number of participants | We have more than 8 UK centres willing to participate in the study. One concern is that recruitment to this study might be difficult, as women might not agree to be randomised to no intervention. As this a pilot study, we plan to recruit 20 women in the first group (13 women in the cerclage group and 7 women in the control group) and 11 women in the second group (7 women in the cerclage group and 4 women in the control group), so 31 participants in total. The rational for choosing randomisation of 2:1 (cerclage:expectant management) is that women often request the cerclage as a treatment in view of the favourable published observational data and the extremely poor outcome in the pregnancies which are expectantly managed. Therefore, participating in the trial has 2 out of 3 chance of receiving the cerclage and 1 out of 3 of being randomised to the expectant management. This pilot trial will provide the data required for a full funding application to the NIHR RFPB programme. |
| | Primary outcome measure(s) Time to delivery (from randomisation to birth). |
| | Secondary outcome measure(s) 1. Gestation at delivery |
| | · · · |
| | Gestation at delivery |
| Cuitouio fou | <ol> <li>Gestation at delivery</li> <li>Preterm birth before 28, 32 and 34 weeks' gestation</li> </ol> |
| Criteria for evaluation | <ol> <li>Gestation at delivery</li> <li>Preterm birth before 28, 32 and 34 weeks' gestation</li> <li>Birthweight</li> </ol> |
| | <ol> <li>Gestation at delivery</li> <li>Preterm birth before 28, 32 and 34 weeks' gestation</li> <li>Birthweight</li> <li>Stillbirth</li> </ol> |
| | <ol> <li>Gestation at delivery</li> <li>Preterm birth before 28, 32 and 34 weeks' gestation</li> <li>Birthweight</li> <li>Stillbirth</li> <li>Neonatal death</li> </ol> |
| | <ol> <li>Gestation at delivery</li> <li>Preterm birth before 28, 32 and 34 weeks' gestation</li> <li>Birthweight</li> <li>Stillbirth</li> <li>Neonatal death</li> <li>Survival to discharge</li> </ol> |

| | 10. Maternal morbidity (defined as thromboembolic complications, chorioamnionitis, urinary tract infection treated with antibiotics, pneumonia, endometritis, eclampsia, HELLP syndrome, death, or any other significant morbidity) |
|---|---|
| | This study is planned to take place in a number of centres in the |
| Sources of funding | UK. The trial is partially funded by the Twins And Mutiple Births Association (TAMBA). |
| Anticipated start date: | March 1 <sup>st</sup> , 2017 |
| Anticipated primary completion date: | December 31 <sup>st</sup> , 2018 |
| Sponsor/Co-Sponsor | Nadia Azzouzi Tel: 02082666488 Fax: 020 8725 0794 Email:nazzouzi@sgul.ac.uk |
| Key Contact names | Sponsor representative: Nadia Azzouzi Tel: 02082666488 Fax: 020 8725 0794 Email:nazzouzi@sgul.ac.uk |
| | Chief Investigator: Dr Asma Khalil<br>Email: akhalil@sgul.ac.uk<br>Tel: 0208 725 0071<br>Fax: +44 20 8725 0079 |

### 4 Background

Preterm birth remains the leading cause of perinatal mortality and morbidity.<sup>1</sup> It is also associated with societal and economic burden, with a substantial risk of long-term mental and physical disability.<sup>1</sup> Twin pregnancies are at increased risk of perinatal mortality and morbidity largely due to preterm birth and complications related to monochorionicity such as twin to twin transfusion syndrome (TTTS).<sup>2-5</sup> Up to 2-3% of births in the UK are from multiple pregnancies and the incidence continues to rise, mainly due to increasing maternal age and the widespread use of assisted reproductive technologies.<sup>2</sup> More than half of twin pregnancies deliver before 37 weeks and approximately 15% have preterm birth prior to 34 weeks' gestation.<sup>2,6</sup> Adverse neonatal outcomes include neonatal death, respiratory and neurological complications, the likelihood of which are related to the gestational age at delivery, ranging from 77% in those born before 28 weeks to less than 2% at term.<sup>7</sup>

Cervical insufficiency, defined as painless second-trimester cervical dilatation, is a well-recognised aetiology of preterm birth. In twin pregnancies measurement of cervical length can be used to predict those at increased risk of spontaneous early preterm delivery.<sup>2,8-10</sup> However, an effective prevention strategy for preterm delivery has yet to be discovered. In singleton pregnancies, progesterone treatment in women identified as being at increased risk of preterm birth was associated with an almost 50% reduction in the incidence of preterm birth before 34 weeks.<sup>11-13</sup> Furthermore, in women at increased risk of (singleton) preterm labour, placement of cervical cerclage when cervical shortening was detected has been associated with a reduction in the risk of preterm birth.<sup>14,15</sup> Unfortunately, however, preventive measures such as bed rest, progesterone therapy and cervical cerclage, have had disappointing results in twin pregnancies.<sup>11,16-19</sup> In fact, bed rest was associated with a significant *increase* in the rate of early preterm delivery. Progesterone therapy and elective cervical cerclage did not reduce the risk significantly.<sup>11,17-20</sup>

In women presenting with an already dilated cervix and/or bulging membranes in the second trimester, the rate of preterm birth has been reported to be as high as 90%, leading to miscarriage, neonatal death or extreme prematurity, and often associated with chorioamnionitis. According to the published observational and limited randomised controlled trials, placement of an emergency cerclage was associated with a longer mean cerclage-to-delivery interval, and lower rates of preterm delivery before 34 weeks and of neonatal morbidity. Therefore, emergency cerclage is likely to be associated with improved perinatal outcome in a cohort of pregnancies with a painless dilated cervix putting them at very high risk of extremely preterm birth. However, most of these studies included singleton pregnancies. In their trial including 11 twin pregnancies, Gupta et al reported that emergency cerclage was associated with a "good outcome", where the pregnancy reached 32 weeks, with a healthy neonate in 36.4% of twin pregnancies. In these studies, predictors of poor outcome included prolapsed membranes, evidence of intra-amniotic or systemic infection, symptomatic presentation, cervical dilatation greater than 3 cm, or gestational age beyond 22 weeks at placement of the cerclage.

There are no randomised clinical trials investigating the role of emergency cerclage solely in multiple pregnancies. Only one randomised study included a very small number of twin pregnancies, along with several singleton pregnancies.<sup>21</sup> This compared a group of 13 women (10 singleton and 3 twin pregnancies) allocated to emergency cerclage with a second group of 10 women (6 singleton and 4 twin pregnancies) who had bed

rest only. This study demonstrated that the cerclage group did significantly better compared with the bed-rest group in mean randomisation-to-delivery interval (54 vs 20 days, P=0.046), preterm delivery before 34 weeks (54% vs 100%, P=0.02), and compound neonatal morbidity, defined as admission to the neonatal intensive care unit and/or neonatal death (62.5% vs 100%; P=0.02; relative risk, 1.6; 95% confidence interval, 1.1-2.3). The main criticism of this study was its very small size. Observational studies in twin pregnancies have reported promising results.<sup>29,30</sup> Levin et al reported the pregnancy outcome in 14 women with twin gestations complicated by cervical shortening/effacement only or bulging membranes through the external os, who underwent emergency cerclage. The average time interval between cerclage placement and delivery was 80.2 days in the group with cervical shortening/effacement, and 48.5 days in the group with bulging membranes.<sup>29</sup> More recently, Aguilera et al reported mean pregnancy prolongation of 60.25 days with 76.9% neonatal survival in a case series of 12 multiple pregnancies with painless cervical dilation and exposed fetal membranes that underwent emergency cerclage. A recent retrospective cohort study has demonstrated that the combination of cerclage, indomethacin, and antibiotics in twin pregnancies with cervix dilated ≥1 cm before 24 weeks was associated with significantly longer latency period from diagnosis to delivery (6.7 weeks; 10.5 vs 3.7 weeks), decreased incidence of spontaneous preterm birth at any given gestational age (52.6% vs 94.7%, 44.7% vs 89.4%, 31.6% vs 89.4% for preterm birth <34 weeks, <32 weeks and <28 weeks' gestation, respectively), and improved perinatal outcome (reduced perinatal mortality 27.6% vs 59.2%, neonatal intensive care unit admission 75.9% vs 97.6%, and composite adverse neonatal outcome 33.9% vs 90.5%) when compared with expectant management.<sup>31</sup> A summary of the studies of cerclage in twin pregnancies with dilated cervix is shown in Table 1.

These results are promising, but these studies are retrospective, include small numbers of pregnancies and are likely to be biased in view of their observational nature and the possibility of selecting less favourable cases for intervention versus conservative management. Moreover, there are risks associated with insertion of an emergency cerclage, such as rupture of the membranes during the procedure, which inevitably is followed by delivery.

Severe TTTS, which affects 10-15% of monochorionic twin pregnancies, is associated with an over 50% risk of delivering before 34 weeks. 32,33 Studies have demonstrated that, in addition to factors predicting fetal survival, such as fetal Doppler or Quintero staging, cervical length is a strong predictor of preterm delivery in pregnancies complicated by TTTS. 33,34 Cervical shortening in TTTS is likely to be mainly because of increased pressure in the amniotic cavity secondary to the severe polyhydramnios. Therefore, it could be argued that in this subgroup of twin pregnancies, emergency cerclage following laser therapy might be an effective intervention in those pregnancies with a short cervix. In fact, an observational study has reported that placement of an emergency cerclage in these pregnancies was associated with prolongation of the pregnancy. In this small study which included 5 pregnancies with a short cervix (<15mm; less than the 5th centile) which were managed expectantly and 9 pregnancies with a short cervix which had emergency cerclage inserted following the Laser surgery, the gestational age at delivery was 23.1 weeks and 30.5 weeks, respectively (p=0.004). Furthermore, there were 16 (89%) and 4 (40%) surviving twins in cases

with and without cerclage, respectively (p=0.01).<sup>34</sup> Despite these promising results, a multicentere, retrospective cohort study including 163 patients with a short cervix (defined as  $\leq$ 25mm) at the time of the Laser surgery for TTTS, reported no difference in the gestational age at delivery (28.8 ± 5.4 vs 29.1 ± 5.6 weeks with and without cerclage, respectively) or perinatal mortality between the group which had cerclage (n=79) and the group which did not (n=84).<sup>37</sup> However, the cerclage was performed more frequently for a cervical length of  $\leq$  15 mm, so this group was at a higher risk of preterm birth and adverse outcome. To date there are no randomised trials investigating the role of emergency cerclage in these high-risk pregnancies.

The study hypothesis is that the placement of an emergency cervical cerclage prolongs the pregnancy in (1) twin pregnancies with a dilated internal cervical os between 14+0 and 26+0 weeks, and (2) in monochorionic twin pregnancies complicated by TTTS treated by Laser surgery between 16+0 and 26+0 weeks' gestation in whom a short cervix (<15mm) is identified.

### 5 Study objectives

### 5.1 Primary objective

The main objective of the study is to investigate whether the insertion of an emergency cerclage will prolong the pregnancy in twin pregnancies in each of the two study groups.

### 5.2 Secondary objectives

Other study objectives include determining the effect of the emergency cerclage on adverse perinatal outcome, defined as preterm birth less than 32 weeks' gestation, a composite outcome of stillbirth, neonatal death, intraventricular haemorrhage, periventricular leukomalacia, respiratory distress syndrome, bronchopulmonary dysplasia, retinopathy of prematurity, necrotising entercolitis, proven neonatal sepsis, or the need for ventilation. We also plan to investigate the length of admission to the neonatal unit and maternal morbidity.

### 6 Trial design

Open-label multi-centre randomised controlled trial.

### 7 Participation selection criteria

There will be no exceptions (waivers) to eligibility criteria prior to participant inclusion into the study. Any questions raised about eligibility should be addressed prior to entering the participant.

The eligibility criteria have been carefully considered and are standards used to ensure the trial results can be appropriately used to make future treatment decisions for other people

with similar disease or medical condition. It is therefore vital that exceptions are not made to the following detailed selection criteria.

All participants that are screened for inclusion into the study must be entered onto the Sponsor screening log JREOLOG0001 and will be assigned a sequential number. Participants will be considered eligible for enrolment into this trial if they fulfil all of the inclusion criteria and none of the exclusion criteria as defined below.

Eligible participants will be entered onto the Sponsors Subject ID log JREOLOG0002 and assigned a Trial specific Identification number in a pre-agreed format in accordance with Site Identifier and next sequential numerical value, e.g. SG001.

#### 7.1 Inclusion criteria

- Twin pregnancies presenting with an open cervix between 14 and 26 weeks, OR
- Monochorionic twin pregnancies complicated by TTTS treated by Laser surgery between 16+0 and 26+0 weeks' gestation in whom a short cervix (<15mm) is identified.
- Age >18 years
- Informed consent

#### 7.2 Exclusion criteria

- Cervical dilatation ≥5cm
- Amniotic membranes prolapsed beyond external os into the vagina, unable to visualise cervical tissue
- Preterm premature rupture of the membranes (PPROM) at the time of diagnosis of dilated cervix
- Major fetal malformations unrelated to TTTS
- Intrauterine death of one or both fetuses
- Symptoms or signs of threatened imminent delivery, e.g. painful regular uterine contractions, active vaginal bleeding, history of ruptured membranes, or suspected chorioamnionitis [based on maternal uterine tenderness, a temperature of 38°C or greater, significant leucocytosis (>15,000 x 10<sup>6</sup>/L) or elevated C-reactive protein (>15 mg/L), or maternal tachycardia].<sup>38</sup>
- Placenta praevia
- Monochorionic monoamniotic twin pregnancies
- Prophylactic cervical cerclage
- Women who are not able to give valid consent, e.g. unconscious or severely ill
- Mental health disorder which impairs the ability to give fully informed consent
- Women under the age of 18 years
- Higher order multiple pregnancies

### 8 Participant Recruitment process

Patient recruitment at a site will commence only once there is evidence that the following approval/essential documents are in place:

- 1. REC approval
- 2. Final sponsorship and host site permissions

All subjects who wish to enter the study will be fully screened and consented by the Chief Investigator or an appropriate delegate.

Patients will be invited to participate in the trial if they have (1) a twin pregnancy and present with an open cervix or (2) a monochorionic twin pregnancy complicated by TTTS treated by Laser surgery, and have a short cervix. These women usually present with an incidental finding of a shortened dilated cervix on cervical length surveillance, or they present with subjective complaints of increased pelvic pressure or vaginal discharge and then undergo cervical length assessment (either ultrasound or speculum examination, or both). Eligible women will be identified by staff in the antenatal clinic, delivery suite, ultrasound department, fetal medicine unit and day assessment unit. All eligible women will be given verbal and written information about the trial and be invited to take part.

The trial will be conducted by the sponsor, participating sites and all investigators in accordance with the protocol, the Declaration of Helsinki, the guidelines on Good Clinical Practice (GCP) and all legal requirements, including applicable national legislation, for the conduct of this trial.

### 9 Study procedures

#### 9.1 Informed consent

It is essential that all trial teams undertaking the informed consent process have signed the Sponsor's Delegation of Responsibilities Log JREOLOG0004 to ensure that the person has been delegated the responsibility by the study CI/PI. All personnel taking informed consent must be GCP trained. Refer to Sponsor SOP JREOSOP0027.

Informed consent will be obtained from eligible women by a member of the research team after confirming the eligibility, inclusion and exclusion criteria.

The Principal Investigator or designee will explain to the patient that she is under no obligation to enter the trial and can withdraw at any time during the trial, without having to give a reason. Those who agree to take part will be asked to sign a Consent Form prior to any study investigation or treatment. The participants' general practitioners will be informed in writing about the trial, and the hospital notes of those receiving an emergency cerclage will be marked with a sticker labelled 'emergency cerclage'. Those who decline to participate in the randomised trial will be asked if they consent to the research team following up their pregnancy outcomes and recording anonymised pregnancy and neonatal outcome data in the study registry. The consent form will allow women to

# specify that they are willing for their data to be collected but prefer not to participate in the randomised controlled study.

A copy of the signed Informed Consent Form (ICF) along with a copy of the most recent approved Patient Information Sheet (PIS) will be given to the study participant. An original signed & dated ICF will be retained in the medical notes and a copy will be placed in the Investigator Site File (ISF). A copy of the signed ICF will also be given to the participant.

If new information results in significant changes to the risk-benefit assessment, the ICF will be reviewed and updated as necessary. All participants, including those already being treated, will be informed of the new information, given a copy of the revised ICF and asked to re-consent if they choose to continue in the study.

### 9.2 Randomisation procedure

Within each of the two study groups, participants will be randomly assigned (2:1) to the 'emergency cerclage' or 'control/expectant management' groups, using a web-based application. Participants and investigators will be aware of the allocation, as masking will be impossible because of the nature of the intervention. At the time of randomisation, the patients will be informed of the possible side-effects of emergency cerclage, such as risk of rupture of the membranes during the procedure.

### 9.3 Discontinuation/withdrawal of participants and stopping rules

In consenting to the trial, participants are consenting to trial treatments, trial follow-up and data collection. However, an individual participant may stop treatment early or be stopped early for any one of the following reasons:

Intercurrent illness that prevents further protocol treatment

Any change in participant's condition that in the investigator's opinion justifies the discontinuation of treatment.

Withdrawal of consent by the participant

As participation in the trial is entirely voluntary, the participant may choose to discontinue participation at any time without penalty or loss of benefits to which she may be entitled. Although not obliged to give a reason for discontinuing her participation, a reasonable effort should be made to establish this reason, whilst remaining fully respectful of the participant's rights. Participants who discontinue study participation for any of the above reasons should remain in the study for the purpose of follow-up and data analysis.

If a participant chooses to discontinue they should be continued to be followed up as closely as possible to the follow-up schedule defined in the protocol, providing they are willing. However, if the participant confirms they do not wish to participate in the scheduled follow-up data collection visits, then data that have already been collected should be kept and analysed according to the ITT principle for all participants who stop follow-up early.

Participants who stop the trial follow-up early will not be replaced.

### 9.4 Participant transfers

If a participant moves from the area making, continued follow-up at their consenting centre inappropriate, every effort should be made for them to be followed up at another sponsor approved trial centre. Written consent should be taken at the new centre and then a copy of the participant's CRF should be provided to the new centre. Responsibility for the participant remains with the original consenting centre until the new consent process is complete.

### 9.5 Lost to Follow-up

For studies conducted in the UK, the NHS number may be used to trace participants who may have changed their GP; specific consent may be required to utilise this.

### 9.6 Definition of the End of Trial

The trial will be completed as soon as 10 patients are included in each of the 4 arms. The End of the Trial is defined as the Last Patient Last Visit (LPLV) or the last data entry point. The REC and the Sponsor will be notified of the end of trial within 90 days of its planned completion or within 15 days if the study is terminated early.

### 10 Study Procedures

### 10.1 Measurement of cervical length

Cervical length will be measured in the usual way (part of the routine care; not considered as a specific study investigation). The woman will be asked to empty her bladder, placed in the lithotomy position, and the transvaginal probe will be placed in the anterior fornix of the vagina. A sagittal view of the cervix will be obtained and the calipers used to measure the distance between the triangular area of echodensity at the external os and the V-shaped notch at the internal os. Each examination will be performed over a period of around three minutes. In around 1% of cases, dynamic cervical changes, due to uterine contractions, are observed. In such cases the shortest measurement will be recorded. Presence or absence of funnelling/cervical dilatation at the internal os will be documented. The researchers will receive appropriate training on measurement of cervical length.

### 10.2 Screening for infections

Women will routinely (not considered as a specific study investigation) have bacteriological investigation. Treatment using the appropriate antibiotic will be given if there is an infection. If they are allocated to the cerclage group, the cerclage will be inserted after completion of the treatment.

An amniocentesis of the presenting twin might be performed, according to local protocols, to quantify amniotic glucose, leucocytes, IL-6 and leucocyte esterase levels and for microbiological film. If the initial assessment (within 24 hours) suggests the presence of infection [positive gram stain/amniotic fluid leucocyte count (≥6 leucocytes per high-power field or >30 cells/mm3) and/or amniotic fluid glucose concentration of ≤15 mg/dL]<sup>39</sup>, women will not be randomised.

#### 10.3 Baseline assessments

The planned baseline assessments include assessment for the inclusion and exclusion criteria and data collection.

### 10.4 Interventions (Insertion of Cerclage)

A McDonald or Shirodkar-type rescue cerclage will be placed. The choice of surgical approach will be at the discretion of the operating clinician and in line with local common practice. The local practice will be clarified during the initial site capacity and capability assessments. The cerclage will be inserted by a competent obstetrician that has performed more than 15 cerclage procedures (including both elective and emergency). Distension of the urinary bladder and/or a Foley balloon will be used when necessary to replace the fetal membranes into the uterine cavity. Participants will be admitted pre-operatively and reevaluated for the previously described exclusion criteria. They will receive peri-operative indomethacin for a period of between 6 and 24 hours. Post-operatively, women can be discharged if there is no uterine activity, rupture of the membranes, symptoms or signs of infection after 24 to 48 hours.

In women aiming for a vaginal birth, the cervical suture will be removed by a simple speculum examination at 35-36 weeks' gestation. If the woman is planning Caesarean section, the suture will be removed at the time of the Caesarean, at the end of the procedure.

However, if at any time rupture of the membranes occurs, or the mother develops symptoms or signs of uterine infection (chorioamnionitis), significant vaginal bleeding or regular painful uterine contractions, the cervical suture should be removed without delay.

If the pregnancy continues without complications, delivery will be planned in line with NICE guidelines (dichorionic twin pregnancy at 37 weeks' gestation and monochorionic twin pregnancy at 36 weeks' gestation).<sup>2</sup> Monochorionic twin pregnancy complicated by TTTS treated by Laser will have planned delivery at 34-36 weeks according to local protocols.

### 10.5 Follow-up visits

Follow-up visits for ultrasound assessment of fetal growth and cervical length will be carried out as per the local protocol (approximately every four weeks in dichorionic diamniotic twin pregnancies and every 2-3 weeks in monochorionic diamniotic twin pregnancies). A course of steroids (two intramuscular injections of betametasone/dexametasone 12 mg, 24 hours apart) will be administered in the week before any planned birth after 23 weeks' gestation.

### 10.6 Data collection

Information on the baseline characteristics of the patients, including demographic data, measurements for calculation of body mass index, and obstetrical and medical histories, will be collected at recruitment and recorded in a computer database. Data on pregnancy outcomes will be obtained from the hospital maternity and neonatal records or the patients' general medical practitioners. The obstetric records of all women who experience preterm birth will be examined to determine whether the delivery was medically indicated or

spontaneous. Spontaneous deliveries will include those with spontaneous onset of labour and those with rupture of membranes before labour. Quality control of the collected data and verification of adherence to protocols at the different centres will be performed on a regular basis by the trial coordinator.

### 10.7 Study flow chart and summary table of study assessments

Please refer to Appendix 1 and Appendix 2.

### 11 Study Timeline

Please refer to Appendix 3.

### 12 Safety Events

#### 12.1 Definitions

Adverse Event (AE)—any untoward medical occurrence in a participant whether it is considered to be related to the intervention or not, that includes a clinical sign, symptom, or condition and/or an observation of a near incident. This does not include pre-existing conditions recorded as such at baseline; continuous persistent disease or a symptom present at baseline that worsens following administration of trial intervention.

**Serious Adverse Event (SAE)** - any Adverse Event or untoward medical occurrence in a trial participant that can be wholly or partly due to the intervention which resulted in any of the following:

- Death
- Is life-threatening (places the participant, in the view of the Investigator, at immediate risk of death)
- Requires hospitalisation or prolongation of existing hospitalisation (hospitalisation is defined as an inpatient admission, regardless of length of stay, even if it is a precautionary measure for observation, including hospitalisation for an elective procedure for a pre-existing condition)
- Results in persistent or significant disability or incapacity (substantial disruption of one's ability to conduct normal life functions)
- Consists of a congenital anomaly or birth defect (in offspring of participants regardless of time of diagnosis)
- Is another important medical condition

Important medical events that may not be immediately life-threatening or result in death or hospitalisation but may jeopardise the participant or require intervention to prevent one of the outcomes listed in the definition of serious AE will also be considered serious.

### 12.2 Recording Adverse Events (AEs)

All Adverse Events will be recorded in the hospital notes in the first instance.

A record of all AEs, whether related or unrelated to the treatment, will also be kept in the CRF and the Sponsor's AE Log JREOLOG0007.

If the Investigator suspects that the disease or condition has progressed faster due to the intervention, then she will report this as an unexpected adverse event to the sponsor.

### 12.3 Investigator Responsibilities relating to Safety Reporting

Collection, recording and reporting of AEs (including serious and non-serious events and reactions) to the Sponsor will be done according to the Sponsor's Safety reporting for non-CTIMP studies SOP JREOSOP0033.

All SAEs will be recorded in the hospital notes and the CRF, and the Sponsor's AE Recording Log JREOLOG0007. The AE Log will be sent to the Sponsor on request and every 2 months.

All SAEs will be reported both to the Sponsor via the JREO & REC using the SAE report form for research other than CTIMPs (non-CTIMPs) published on the HRA website.

The Chief or Principal Investigator, or a member of the research team, at any participating site will complete the SAE form which will be faxed both to the JREO on 020 8725 0794 or E-mailed to <a href="maileographe-adverseevents@sgul.ac.uk">adverseevents@sgul.ac.uk</a>, within 48hrs of the Investigator becoming aware of the event, and via email to the relevant REC.

The Chief or Principal Investigator will respond to any SAE queries raised by the Sponsor as soon as possible. Follow-up reports must continually be completed within an acceptable time-frame and sent as detailed above until the reportable event is considered resolved.

Events will be followed up until resolution; any appropriate follow-up information will be clearly marked as such and reported to the sponsor via the JREO as above in a timely manner.

Full reports should be completed and submitted to REC within 15 days of the event.

### 12.4 Notification of deaths

Only deaths that are assessed to be caused by the trial intervention will be reported to the Sponsor. This report will be immediate.

### 13 Data management and quality assurance

### 13.1 Confidentiality

All data will be handled in accordance with the Data Protection Act 1998.

The Case Report Forms (CRFs) will not bear the participant's name or other directly identifiable data. The participant's trial Identification Number (ID) only will be used for identification. The sponsor Subject ID log JREOLOG0002 can be used to cross reference participants' identifiable information.

#### 13.2 Data collection tool

Case Report Forms will be designed by the CI. All data will be entered legibly in black ink with a ball-point pen. If the Investigator makes an error, it will be crossed through with a single line in such a way as to ensure that the original entry can still be read. The correct entry will then be clearly inserted. The amendment will be initialled and dated immediately by the person making the correction. Overwriting or use of correction fluid will not be permitted.

It is the Investigator's responsibility to ensure the accuracy of all data entered and recorded in the CRFs. The Staff Delegation of Responsibilities Log JREOLOG0004 will identify all trial personnel responsible for data collection, entry, handling and managing the database.

### 13.3 Incidental Findings

All subjects will be informed in a timely manner, both verbally and in writing, of any new information, findings or changes to the way the research will be conducted that are of potential relevance for participants or their families and might influence their willingness to continue in this study.

### 13.4 Data handling and analysis

The trial will use an online secure database. Quality Control will be applied at each stage of data handling to ensure that all data are reliable and have been processed correctly.

### 14 Archiving arrangements

The trial essential documents along with the trial database will be archived in accordance with the sponsor SOP JREOSOP0016. The agreed archiving period for this trial will be 10 years.

### 15 Statistical design

### 15.1 Endpoints

### 15.1.1 Primary endpoints

Time to delivery (from randomisation to birth).

### 15.1.2 Secondary endpoints

- Gestation at delivery
- Preterm birth before 28, 32 and 34 weeks' gestation
- Birthweight
- Stillbirth
- Neonatal death
- Survival to discharge

- Days of admission to the neonatal intensive care unit
- Composite outcome of stillbirth, neonatal death, intraventricular haemorrhage<sup>40</sup>, periventricular leukomalacia, respiratory distress syndrome, bronchopulmonary dysplasia, retinopathy of prematurity<sup>41</sup>, necrotising entercolitis<sup>42</sup>, proven neonatal sepsis, or the need for ventilation
- Days of maternal admission for preterm labour
- Maternal morbidity (defined as thromboembolic complications, chorioamnionitis, urinary tract infection treated with antibiotics, pneumonia, endometritis, eclampsia, HELLP syndrome, death, or any other significant morbidity)

### 15.2 Sample size calculation

### Study 1: Twin pregnancies presenting with an open cervix Group

We performed a sample size calculation based on the GA and preterm birth percentage (45% and 99% for with and without cerclage). Also included the outputs based on the preterm birth percentage of 45% and 95% for with and without cerclage.

An experiment with 6 women in the cerclage group and 3 women in the control group will have 80% power to detect the gestational age (at delivery) difference of 6 weeks or greater between cerclage and control groups at a significance level of 5%. Assuming the percentage of preterm birth at less than 32 weeks for the cerclage and control groups as 45% and 99%, respectively, an experiment with 15 women in the cerclage group and 8 women in the control group will achieve 80% power with the statistical significance of 5%. With the assumption that approximately 14 births occurring among these women in less than 32 weeks, an experiment with 20 women will also detect a hazard ratio of 0.34 or less in favour of the cerclage group - the cerclage group will be 66% less likely to give a birth at any time point before 32 weeks compared with the control group - with at least 80% power. These calculations do not include the loss to follow-up which should be considered by including one additional subject in each group.

Preterm birth percentage:

Cerclage group = 45%

Control group = 95%

Sample size:

Cerclage group = 19

Control group = 10

HR = 0.39

# Study 2: Monochorionic Twin pregnancies complicated by TTTS treated by Laser surgery with short cervix (<15mm) Group

We have more than 8 UK centres willing to participate in the study. One concern is that recruitment to this study might be difficult, as women might not agree to be randomised

to no intervention. As this a pilot study, we plan to recruit 20 women in the Study 1 (13 women in the cerclage group and 7 women in the control group) and 11 women in the second Study 2 (7 women in the cerclage group and 4 women in the control group), so 31 participants in total. The rational for choosing randomisation of 2:1 (cerclage:expectant management) is that women often request the cerclage as a treatment in view of the favourable published observational data and the extremely poor outcome in the pregnancies which are expectantly managed. Therefore, participating in the trial has 2 out of 3 chance of receiving the cerclage and 1 out of 3 of being randomised to the expectant management.

An experiment with 13 women in the cerclage group and 7 women in the control group in the Study 1 will have 80% power to detect the gestational age (at delivery) difference of 6 weeks or greater between cerclage and control groups at a significance level of 5%. Similarly, an experiment with 7 women in the cerclage group and 4 women in the control group in the Study 2 will have 80% power to detect the gestational age (at delivery) difference of 6 weeks or greater between cerclage and control groups at a significance level of 5%. These calculations include the 5% loss to follow-up by including one additional subject in each group. The above calculations also assume that the between centre variability is negligible for the outcome of interest. This pilot trial will provide the data required for a full funding application to the NIHR RFPB programme.

### 15.3 Statistical analysis plan

Statistical analyses will be performed according to intention to treat. The primary analysis will compare the time to delivery (from randomisation to birth) in weeks. Other outcomes, such as gestational age at delivery, preterm birth before 28, 32 and 34 weeks' gestation, median birthweight, stillbirth, neonatal death and survival to discharge will be compared between the 2 arms of each study group as secondary outcomes. A number of statistical tests, including Pearson's chi-squared test [RR, (95%Cls)], Logrank test [HR, (95%Cls)] and 2-sample student's t-test [mean  $\pm$  SD], will be used to analyse the various outcomes.

### 16 Ethics and Research Governance requirements

Before any site can enrol patients into the trial, the Principal Investigator must ensure that written permission to proceed has been granted by that Trust Research & Development (R&D). The site must conduct the trial in compliance with the protocol as agreed by the Sponsor and which was accepted by the Research Ethics Committee (REC).

The Chief Investigator will be provided (via the Sponsor) with file indices, e.g. JREODOC0003 TMF index and JREODOC0004 ISF index, for use with SOP JREOSOP0019 'Preparation and Maintenance of the TMF'. The CI will be responsible for the maintenance of the TMF and may delegate the responsibility of ISF file maintenance to the PI at each participating site.

It is the responsibility of the PI at each site to ensure that all subsequent amendments gain the necessary approval. Refer to JREOSOP0011 'Management of Amendments'.

Within 90 days after the end of the trial, the CI and Sponsor will ensure that the REC is notified that the trial has finished. If the trial is terminated prematurely, those reports will be made within 15 days after the end of the trial. Refer to JREOSOP0015 'End of study declaration'.

The CI will supply an End of Study report of the clinical trial to the REC within one year after the end of the trial. The sponsor can provide JREODOC0059 End of study Report template.

### 16.1 Annual Progress Reports (APRs)

The Chief Investigator will prepare the APR in accordance with JREOSOP0043. Following review by the sponsor the report will be sent to the REC. The APR is due for submission annually within 30 days of the anniversary date on which the favourable opinion was given by the Ethics committee, until the trial is declared ended.

### 16.2 Notification of Serious Breaches of GCP and/or the protocol

Any Protocol Deviations or Violations will be documented using JREODOC0061, and entered onto the Sponsor's log JREOLOG0005. Potential Serious Breaches and Urgent Safety Measures will be recorded both on the Sponsor's Log JREOLOG0005 and processed according to JREOSOP0012 and where necessary JREOSOP0032.

A "serious breach" is a breach which is likely to affect to a significant degree:

- (a) The safety or physical or mental integrity of the participants of the trial; or
- (b) The scientific value of the trial.

The CI will notify the Sponsor immediately of any case where there is a possible serious breach.

#### 16.3 Direct access to source data

The Investigator(s)/institution(s) will permit trial-related monitoring, audits, REC review, and regulatory inspection(s), providing direct access to source data/documents. Trial participants are informed of this during the informed consent discussion. Participants will consent to provide access to their medical notes.

### 17 Finance

The trial is partially funded by the Twins and Multiple Births Association (TAMBA), which is the largest UK charity providing support to multiple pregnancies. The funding will contribute to the salary of a research midwife who will coordinate the trial.

### 18 Insurance and indemnity

NHS bodies are liable for clinical negligence and other negligent harm to individuals covered by their duty of care. NHS Institutions employing researchers are liable for negligent harm caused by the design of studies they initiate.

### 19 Development policy

The sponsor, participating sites and all investigators involved in the study shall treat all information and data related to the study as confidential and with the proper respect for the privacy of each participant. The parties shall equally warrant to not disclose such information to third parties or disclose such publicly, but shall use such information solely for the purpose of this study. All data shall be coded or de-identified prior to transfer of such data to sponsor.

Parties have expressly agreed that any and all data collected and prepared in the context of the study shall be the property of the sponsor, provided that the participating sites shall remain the owner of their source data and may utilise such data as it deems appropriate without the approval of sponsor.

The participating sites and their proper investigators warrant that they shall not perform the study without having obtained the proper, written informed consent from each participant, in accordance with applicable legislation and as approved by the appropriate ethics committee/review board.

### 20 Publication policy

Publication: "Any activity that discloses, outside of the circle of trial investigators, any final or interim data or results of the Trial, or any details of the Trial methodology that have not been made public by the Sponsor including, for example, presentations at symposia, national or regional professional meetings, publications in journals, theses or dissertations."

All scientific contributors to the Trial have a responsibility to ensure that results of scientific interest arising from Trial are appropriately published and disseminated. The Sponsor has a firm commitment to publish the results of the Trial in a transparent and unbiased manner without consideration to commercial objectives.

To maximise the impact and scientific validity of the Trial, data shall be consolidated over the duration of the trial, reviewed internally among all investigators and not be submitted for publication prematurely.

### 20.1 Before the official completion of the Trial

All publications during this period are subject to permission by the Sponsor. If an investigator wishes to publish a sub-set of data without permission of the Sponsor during this period, the steering committee shall have the final say.

### 20.2 Up to 180 days after the official completion of the Trial

During this period the Chief Investigator shall liaise with all investigators and strive to consolidate data and results, then submit a manuscript for peer review with a view to publication in a reputable academic journal or similar outlet as the Main Publication.

- The Chief Investigator shall be senior and corresponding author of the Main Publication.
- Insofar as is compatible with the policies of the publication outlet and good academic practice, the other Investigators shall be listed in alphabetic order.
- Providers of analytical or technical services shall be acknowledged, but will be listed
  as co-authors only if their services were provided in a non-routine manner as part of
  a scientific collaboration.
- Members of the Steering Group shall be acknowledged as co-authors only if they also contributed in other capacities.
- If there are disagreements about the substance, content, style, conclusions, or author list of the Main Publication, the Chief Investigator shall ask the Steering Group to arbitrate.

### 20.3 Beyond 180 days after the official completion of the Trial

After the Main Publication or after 180 days from Trial end date, any Investigator or group of investigators may prepare further publications. In order to ensure that the Sponsor will be able to make comments and suggestions where pertinent, material for public dissemination will be submitted to the Sponsor for review at least sixty (60) days prior to submission for publication, public dissemination, or review by a publication committee. Sponsor's reasonable comments shall be reflected. All publications related to the Trial shall credit the Chief and Co-Investigators as co-authors where this would be in accordance with normal academic practice and shall acknowledge the Sponsor and the Funders.

### 21 Statement of Compliance

The trial will be conducted in compliance with the protocol, Sponsor's Standard Operating Procedures (SOPs), GCP and the applicable regulatory requirement(s).

The study conduct shall comply with all relevant laws of the EU if directly applicable or of direct effect and all relevant laws and statutes of the country in which the study site is located, including but not limited to the Human Rights Act 1998, the Data Protection Act 1998, the Human Medicines Regulations 2012, ICH GCP, the World Medical Association Declaration of Helsinki entitled 'Ethical Principles for Medical Research Involving Human Subjects' (2008 Version), the NHS Research Governance Framework for Health and Social Care (Version 2, April 2005).

This study will be conducted in compliance with the protocol approved by the REC and according to GCP standards. No deviation from the protocol will be implemented without the prior review and approval of the Sponsor and REC except where it may be necessary to eliminate an immediate hazard to a research subject. In such case, the deviation will be reported to the Sponsor and REC as soon as possible.

### 22 List of Protocol appendices

**Appendix 1** Study flow chart

Appendix 2 Summary table of study assessments

**Appendix 3** Timeline of the proposed pilot study

**Appendix 4** Protocol Amendment/Revision History (chronological order) or a statement "There are currently no amendments"

### 23 References

- 1. Goldenberg RL, Culhane JF, Iams JD, Romero R. Epidemiology and causes of preterm birth. Lancet 2008;371:75–84.
- 2. Visintin C, Mugglestone MA, James D, Kilby MD; Guideline Development Group. Antenatal care for twin and triplet pregnancies: summary of NICE guidance. *BMJ* 2011; **343**: d5714.
- 3. Miller J, Chauhan SP, Abuhamad AZ. Discordant twins: diagnosis, evaluation and management. *Am J Obstet Gynecol* 2012; **206**: 10-20.
- 4. D'Antonio F, Khalil A, Dias T, Thilaganathan B; Southwest Thames Obstetric Research Collaborative (STORK). Weight discordance and perinatal mortality in twins: analysis of the Southwest Thames Obstetric Research Collaborative (STORK) multiple pregnancy cohort. *Ultrasound Obstet Gynecol* 2013; **41**: 643-648.
- 5. D'Antonio F, Khalil A, Dias T, Thilaganathan B; Southwest Thames Obstetric Research Collaborative (STORK). Early fetal loss in monochorionic and dichorionic twin pregnancies: analysis of the Southwest Thames Obstetric Research Collaborative (STORK) multiple pregnancy cohort. *Ultrasound Obstet Gynecol* 2013; **41**: 632-636.
- 6. Souka AP, Heath V, Flint S, Sevastopoulou I, Nicolaides KH. Cervical length at 23 weeks in twins in predicting spontaneous preterm delivery. Obstet Gynecol 1999;94:450-454.
- 7. Guinn DA, Atkinson MW, Sullivan L, Lee M, MacGregor S, Parilla BV, et al. Single vs weekly courses of antenatal corticosteroids for women at risk of preterm delivery: A randomized controlled trial. JAMA. 2001;286:1581–7.
- 8. Skentou C, Souka AP, To MS, Liao AW, Nicolaides KH. Prediction of preterm delivery in twins by cervical assessment at 23 weeks. Ultrasound Obstet Gynecol 2001;17:7-10.

- 9. To MS, Fonseca EB, Molina FS, Cacho AM, Nicolaides KH. Maternal characteristics and cervical length in the prediction of spontaneous early preterm delivery in twins. Am J Obstet Gynecol 2006;194:1360-1365.
- 10. Conde-Agudelo Α, Romero R, Hassan SS, Yeo L. Transvaginal sonographic cervical length for the prediction preterm birth of spontaneous in twin pregnancies: a systematic review and metaanalysis. Am J Obstet Gynecol 2010;203:128.e1-12.
- 11. Romero R, Nicolaides K, Conde-Agudelo A, Tabor A, O'Brien JM, Cetingoz E, Da Fonseca E, Creasy GW, Klein K, Rode L, Soma-Pillay P, Fusey S, Cam C, Alfirevic Z, Hassan SS. Vaginal progesterone in women with an asymptomatic sonographic short cervix in the midtrimester decreases preterm delivery and neonatal morbidity: a systematic review and metaanalysis of individual patient data. Am J Obstet Gynecol 2012;206:124.e1-19.
- 12. Hassan SS, Romero R, Vidyadhari D, Fusey S, Baxter JK, Khandelwal M, Vijayaraghavan J, Trivedi Y, Soma-Pillay P, Sambarey P, Dayal A, Potapov V, O'Brien J, Astakhov V, Yuzko O, Kinzler W, Dattel B, Sehdev H, Mazheika L, Manchulenko D, Gervasi MT, Sullivan L, Conde-Agudelo A, Phillips JA, Creasy GW; PREGNANT Trial. Vaginal progesterone reduces the rate of preterm birth in women with a sonographic short cervix: a multicenter, randomized, double-blind, placebo-controlled trial. Ultrasound Obstet Gynecol 2011;38:18-31.
- 13. Fonseca EB, Celik E, Parra M, Singh M, Nicolaides KH; Fetal Medicine Foundation Second Trimester Screening Group. Progesterone and the risk of preterm birth among women with a short cervix. N Engl J Med 2007;357:462-469.
- 14. Berghella V, Rafael TJ, Szychowski JM, Rust OA, Owen J. Cerclage for short cervix on ultrasonography in women with singleton gestations and previous preterm birth: a meta-analysis. Obstet Gynecol 2011;117:663–671.
- 15. Althuisius SM, Dekker GA, Hummel P, Bekedam DJ, van Geijn HP. Final results of the Cervical Incompetence Prevention Randomized Cerclage Trial (CIPRACT): therapeutic cerclage with bed rest versus bed rest alone. Am J Obstet Gynecol 2001;185:1106–1112.
- 16. Crowther CA, Neilson JP, Verkuyl DA, Bannerman C, Ashurst HM. Preterm labour in twin pregnancies: can it be prevented by hospital admission? BJOG 1989;96:850-853.
- 17. Roman AS, Saltzman DH, Fox N, Klauser CK, Istwan N, Rhea D, Rebarber A. Prophylactic cerclage in the management of twin pregnancies. Am J Perinatol 2013;30:751-754.
- 18. Senat MV, Porcher R, Winer N, Vayssière C, Deruelle P, Capelle M, Bretelle F, Perrotin F, Laurent Y, Connan L, Langer B, Mantel A, Azimi S, Rozenberg P; Groupe de Recherche en Obstétrique et Gynécologie. Prevention of preterm delivery by 17 alphahydroxyprogesterone caproate in asymptomatic twin pregnancies with a short cervix: a randomized controlled trial. Am J Obstet Gynecol 2013;208:194.e1-8.
- 19. Norman JE1, Mackenzie F, Owen P, Mactier H, Hanretty K, Cooper S, Calder A, Mires G, Danielian P, Sturgiss S, MacLennan G, Tydeman G, Thornton S, Martin B, Thornton JG, Neilson JP, Norrie J. Progesterone for the prevention of preterm birth in twin pregnancy (STOPPIT): a randomised, double-blind, placebo-controlled study and meta-analysis. Lancet. 2009;373(9680):2034-2040.

- Rafael TJ, Berghella V, Alfirevic Z. Cervical stitch (cerclage) for preventing preterm birth in multiple pregnancy. Cochrane Database Syst Rev. 2014 Sep 10;9:CD009166. doi: 10.1002/14651858.CD009166.pub2.
- 21. Althuisius SM, Dekker GA, Hummel P, van Geijn HP; Cervical incompetence prevention randomized cerclage trial. Cervical incompetence prevention randomized cerclage trial: emergency cerclage with bed rest versus bed rest alone. Am J Obstet Gynecol 2003;189:907–910.
- 22. Pereira L, Cotter A, Gómez R, et al. Expectant management compared with physical examination-indicated cerclage (EMPEC) in selected women with a dilated cervix at 14(0/7)-25(6/7) weeks: results from the EM-PEC international cohort study. Am J Obstet Gynecol 2007;197:483, e1–e8
- 23. Stupin JH, David M, Siedentopf JP, Dudenhausen JW. Emergency cerclage versus bed rest for amniotic sac prolapse before 27 gestational weeks. A retrospective, comparative study of 161 women. Eur J Obstet Gynecol Reprod Biol 2008;139:32–37
- 24. Ventolini G, Genrich TJ, Roth J, Neiger R. Pregnancy outcome after placement of "rescue" Shirodkar cerclage. J Perinatol 2009;29:276–279
- 25. Daskalakis G, Papantoniou N, Mesogitis S, Antsaklis A. Management of cervical insufficiency and bulging fetal membranes. Obstet Gynecol 2006;107(2 Pt 1):221–226
- 26. Namouz S, Porat S, Okun N, Windrim R, Farine D. Emergency cerclage: literature review. Obstet Gynecol Surv 2013;68:379-88.
- 27. Gupta M, Emary K, Impey L. Emergency cervical cerclage: predictors of success. J Matern Fetal Neonatal Med 2010;23:670–674
- 28. Diago Almela VJ, Martínez-Varea A, Perales-Puchalt A, Alonso-Díaz R, Perales A. Good prognosis of cerclage in cases of cervical insufficiency when intra-amniotic inflammation/infection is ruled out. J Matern Fetal Neonatal Med 2014:1-6. [Epub ahead of print]
- 29. Levin I, Salzer L, Maslovitz S, Avni A, Lessing JB, Groutz A, Almog B. Outcomes of midtrimester emergency cerclage in twin pregnancies. Fetal Diagn Ther 2012;32:246-50.
- 30. Aguilera M, Ramin K, Nguyen R, Giacobbe L, Swartout J. Emergency cerclage placement in multifetal pregnancies with a dilated cervix and exposed membranes: case series. AJP Rep 2013;3:1-4.
- 31. Roman A, Rochelson B, Martinelli P, Saccone G, Harris K, Zork N, Spiel M, O'Brien K, Calluzzo I, Palomares K, Rosen T, Berghella V, Fleischer A. Cerclage in twin pregnancy with dilated cervix between 16 to 24 weeks of gestation: retrospective cohort study. Am J Obstet Gynecol 2016;215:98.e1-98.e11
- 32. Senat MV, Deprest J, Boulvain M, et al. 2004. Endoscopic laser surgery versus serial amnioreduction for severe twin-to-twin transfusion syndrome. N Engl J Med 351: 136–44.
- 33. Robyr R, Boulvain M, Lewi L, et al. 2005. Cervical length as a prognostic factor for preterm delivery in twin-to-twin transfusion syndrome treated by fetoscopic laser coagulation of chorionic plate anastomoses. Ultrasound Obstet Gynecol 25: 37–41.
- 34. Salomon LJ, Nasr B, Nizard J, Bernard JP, Essaoui M, Bussieres L, Ville Y. Emergency cerclage in cases of twin-to-twin transfusion syndrome with a short cervix at the time of surgery and relationship to perinatal outcome. Prenat Diagn 2008;28:1256-61.
- 35. Saunders NJ, Snijders RJ, Nicolaides KH. 1992. Therapeutic amniocentesis in twin-twin transfusion syndrome appearing in the second trimester of pregnancy. Am J Obstet Gynecol 166: 820–4.
- 36. Ville Y, Sideris I, Nicolaides KH 1996. Amniotic fluid pressure in twin-to-twin transfusion syndrome: an objective prognostic factor. Fetal Diagn Ther 11: 176–80.
- 37. Papanna R, Habli M, Baschat AA, Bebbington M, Mann LK, Johnson A, Ryan G, Walker M, Lewis D, Harman C, Crombleholme T, Moise KJ Jr. Cerclage for cervical shortening

- at fetoscopic laser photocoagulation in twin-twin transfusion syndrome. Am J Obstet Gynecol 2012;206:425.e1-7.
- 38. Greenberg MB, Anderson BL, Schulkin J, Norton ME, Aziz N. A first look at chorioamnionitis management practice variation among US obstetricians. Infect Dis Obstet Gynecol 2012;2012:628362.
- 39. Romero R, Yoon BH, Mazor M, et al. A comparative study of the diagnostic performance of amniotic fluid glucose, white blood cell count, interleukin-6, and Gram stain in the detection of microbial invasion in patients with preterm premature rupture of membranes. Am J Obstet Gynecol 1993;169:839-51.
- 40. Papile LA, Burstein J, Burstein R, Koffl er H. Incidence and evolution of subependymal and intraventricular hemorrhage: a study of infants with birth weights less than 1,500 gm. J Pediatr 1978; 92: 529–34.
- 41. International Committee for the Classification of Retinopathy of Prematurity. The International Classification of Retinopathy of Prematurity revisited. Arch Ophthalmol 2005;123:991-9.
- 42. Bell MJ, Ternberg JL, Feigin RD, et al. Neonatal necrotizing enterocolitis: therapeutic decisions based upon clinical staging. Ann Surg 1978; 187: 1–7.

Table 1. Summary of studies on cerclage in twin pregnancy with dilated cervix.

| First<br>author and<br>year | Study<br>design | Cerclage | Controls<br>(no<br>cerclage) | GA | Amniocentesis | Antibiotics | Tocolysis | Time<br>interval<br>until<br>delivery<br>(days) | PTB <28<br>weeks | PTB<br><32<br>weeks | PTB<br><34<br>weeks | PPROM | Neonatal<br>survival |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Althuisius | | | | | | | | | | | | | |
| 2003 | RCT | 3 | 4 | <27 | No | No | No | No data | No data | No data | No data | No data | No data |
| | | | Not | 21.4±2. | | | | | | | | | |
| Parilla 2003 | RC | 11 | specified | 2 | No | N/A | N/A | No data | No data | No data | No data | No data | No data |
| | | | | | | Yes, not | Yes, not | | | | | | |
| Gupta 2010 | RC | 11 | 0 | <27 | No | specified | specified | No data | No data | No data | No data | No data | No data |
| | | | | 20.1±2. | | | | | 2 | | | | 16/20 |
| Levin 2012 | RC | 14 | 0 | 5 | No | All | No | 71.1±44.6 | (14.3%) | N/A | N/A | 2 (14.3) | (80%) |
| Rebarber | | | | | | | | 92 | 2 | | 7 | 2 | 20/24 |
| 2013 | RC | 12 | 0 | 14-23.8 | 12 (100%) | 12 (100) | 12 (100) | (26-145) | (16.6%) | 3 (25%) | (58.3%) | (16.6%) | (83%) |
| Zanardini | | | | | | | | | | | | | 24/28 |
| 20131 | RC | 14 | 0 | 16-26 | No | 14 (100) | 14 (100) | 69 (2-125) | 3 (21%) | 7 (50%) | 7 (50%) | 4 (29%) | (86%) |
| | | | | | Not routinely | | | , | 35 | 54 | , | 35 | , |
| Miller 2014 | RC | 104 | 0 | 16-23.8 | used | 56 (54.3) | 69 (57.3) | 69 (21-99) | (33.7%) | (51.9%) | N/A | (33.7%) | No data |
| Barnabeu | | | | 19.6±4. | | , , | 1 ` ′ | , , | <u> </u> | <b></b> | 3 | 1 | 14/14 |
| 2015 | RC | 7 | 0 | 0 | 7 (100%) | 7 (100) | 7 (100) | 12.1 (4-16) | 2 (28%) | No data | (42.8%) | (14.2%) | (100%) |
| Roman | | | | | , , | , , | , , | , , | 12 | 17 | 20(52.6 | , , | 50/76 |
| 2016 | RC | 38 | 38 | 16-24 | 30 (79%) | 36 (94%) | 29 (76%) | 73±39 | (31.6%) | (44.7%) | %)` | 8 (21%) | (65.8) |

RCT: randomised controlled trial; RC: retrospective cohort; GA: gestational age in weeks; PTB: preterm birth; PPROM: preterm pre-labour rupture of membranes.

### Appendix 1

### Study flow chart



# **Appendix 2.** Summary table of study assessments.

| Study Procedures | Screening | Treatment | Follow-up<br>(neonatal<br>discharge) |
|---|---|---|---|
| Informed consent | √ | | |
| Inclusion/exclusion criteria | $\checkmark$ | | |
| Data collection | <b>V</b> | | |
| Demographics | <b>√</b> | | |
| Baseline | V | | |
| Screening | | | |
| Ultrasound | √ | | |
| Intervention | | √ | |
| Data collection/Telephone call | | | √ |

| ENCIRCLE - trial Protocol V 1.7, 15 <sup>th</sup> May 2018 R&D Protocol Code Number: 17.0004 |
|---|

## Appendix 3. Timeline of the proposed pilot study

| Calendar year | 2017 | | | | | | | | | | 2018 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Calendar month | March | April | May | June | July | August | Sept | Oct | Nov | Dec | Jan | Feb |
| Ethics approval | | | | | | | | | | | | |
| Database design | | | | | | | | | | | | |
| Project set-up | | | | | | | | | | | | |
| Co-ordination among the participating centres | | | | | | | | | | | | |
| Recruitment | | | | | | | | | | | | |
| Data collection | | | | | | | | | | | | |
| Preliminary data analysis, literature review for a peer-reviewed paper | | | | | | | | | | | | |
| Statistical analysis | | | | | | | | | | | | |
| Writing and submission of a peer-reviewed paper and report to the funder | | | | | | | | | | | | |

# Appendix 4

Protocol amendment /Revision History

| Protocol Version and Date | New text |
|---------------------------|----------|